CLINICAL TRIAL: NCT03057613
Title: A Phase II Study of the Addition of Pembrolizumab to Postoperative Radiotherapy in Resected High Risk Cutaneous Squamous Cell Cancer of the Head and Neck
Brief Title: The Addition of Pembrolizumab to Postoperative Radiotherapy in Cutaneous Squamous Cell Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6316
Record Dates: First submitted 2017-02-14; First posted 2017-02-20 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: radiation; resected
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + post operative radiotherapy (Experimental): IMRT 60-66Gy for 6 weeks in combination with Pembrolizumab every 3 weeks for 16 weeks
  Interventions: Drug: Pembrolizumab; Radiation: IMRT 60-66Gy

INTERVENTIONS:
Drug: Pembrolizumab — 200mg every 3 weeks for 16 weeks given by IV infusion
Radiation: IMRT 60-66Gy — 60-66Gy for 6 weeks

SUMMARY:
A small group of skin cancers of the head and neck, called resected cutaneous squamous carcinomas, are more aggressive than most cancers of this type, even after being treated with standard therapy. This trial will use stronger treatment to look at the safety and effectiveness (efficacy) of combining a drug called Pembrolizumab with radiation after a cancer has already been treated to suppress secondary tumor formation in high risk cutaneous squamous cell cancer of the head and neck.

Primary Objective To assess safety by looking at the people with dose limiting responses

DETAILED DESCRIPTION:
Primary Objective:

To assess safety and estimate 1-year progression-free survival (PFS) of postoperative radiation therapy (RT) + concurrent and adjuvant Pembrolizumab in high risk resected cutaneous squamous cell cancer of the head and neck (cSCC-HN).

Secondary Objectives

1. To evaluate the relationship of baseline programmed death-ligand 1 (PD-L1) expression by tumor and tumor-infiltrating lymphocytes (TILs) to preliminary efficacy .
2. To phenotype tumor infiltrating lymphocytes and peripheral blood lymphocytes (PBLs), and investigate tumor suppressor populations including Tregs, myeloid-derived suppressor cells (MDSCs) and cluster of differentiation 8 (CD8) suppressor cells and assess ex vivo for effector function by cytokine production and cytotoxicity assays as well as suppressor function in assays with autologous PBLs.
3. To evaluate the tumor microenvironment (TME), and immune markers at the invasive margin of the tumor, including CD8, PD-1, PD-L1, TIM-3, galectin-9 or HMGB-1, BTLA and HVEM, as well as Lag-3, CTLA-4 and others.
4. To evaluate the genomic and/or transcriptomic profile of these tumors using RNA-seq /Whole Transcriptome Shotgun Sequencing

Trial Design:

This is a phase II trial evaluating the addition of concurrent and adjuvant fixed-dose pembrolizumab in combination with standard intensity-modulated radiation therapy (IMRT), in order to establish safety and estimate efficacy of this regimen to be tested in a subsequent randomized registration trial.

Thirty seven patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of cutaneous squamous cell carcinoma of the head and neck that has been resected with no evidence of gross residual disease (margin positivity is acceptable)
* Patients must have undergone resection of the disease and demonstrate high risk pathologic features including:

  * T4
  * Node positive disease
  * T2/T3N0 disease with any 1 additional feature, including:

    * Recurrent Disease
    * Perineural invasion
    * Lymphovascular space invasion
    * Poorly differentiated histology
    * Positive Margins
    * Satellitosis or in-transit metastases
* Patients are required to have computerized tomography (CT) neck and chest or positron emission tomography/computerized tomography (PET/CT) and have no documented evidence of distant metastases
* Patients must not have a history of the following immunosuppressive conditions:bone marrow transplantation and/or organ transplants and/or chronic rheumatic conditions that require active immunosuppressive therapy. Patients with a history of chronic lymphoid or leukemic malignancies which are not under active therapy (no active therapy within the last 3 months) will be eligible. Patients with chronic lymphoid or leukemic malignancies are eligible with or without active disease as long as they have not had treatment within the past three months.
* Patients may not have had prior therapy with a checkpoint inhibitor (e.g. anti-CTLA-4, anti-PD-1 or anti-PD-L1 therapy)
* Patients may not have had prior radiotherapy (>30Gy) to the area requiring treatment that would result in any overlap of tissue in both fields
* Patients may have received chemotherapy or radiation for a previous, curatively treated malignancy provided at least 2 years have elapsed and there is no current evidence of disease (patients with previous or concurrent additional skin cancers are eligible)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Patients must have adequate laboratory values

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9g/dL or ≥5.6mmol/L without transfusion
  * Serum creatinine ≤ 1.5 times upper limit of normal (ULN) or measured creatinine clearance ≥60mL/min for subject with creatinine levels >1.5 times institutional ULN
  * Serum bilirubin ≤ 1.5 times ULN or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * Aspartate aminotransferase (AST (SGOT)) and alanine aminotransferase (ALT (SPGT)) ≤ 2.5 times ULN or ≤ 5 times ULN for subjects with liver metastases
  * Albumin ≥ 2.5mg/dL

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a known history of active Bacillus Tuberculosis (TB)
* Hypersensitivity to pembrolizumab.
* Has a history of the following immunosuppressive conditions: bone marrow transplantation, and/or organ transplants and/or chronic rheumatic conditions that require active immunosuppressive therapy. Patients with chronic lymphoid/leukemic malignancies that have undergone treatment in the last 3 months will be ineligible.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e.≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiotherapy within 2 weeks prior to study Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or a separate primary squamous cell carcinoma of the skin or a separate primary squamous cell carcinoma of the skin. Patients with chronic lymphoid or leukemic malignancies are eligible with or without active disease as long as they have not had treatment within the past three months.
* Has metastatic disease.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Koyfman, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab + Post Operative Radiotherapy
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who went on study
Arm/Group | Pembrolizumab + Post Operative Radiotherapy
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  60-69 years | 6
  70-79 years | 10
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities
Description: There will be an initial safety run in cohort consisting of an initial safety run in cohort consisting of eight patients to allow for at least six evaluable patients for dose limiting toxicities (DLTs) by the week 20 visit. If a total of 0-2 of the initial six evaluable patients experience DLTs, the safety run in will have been deemed successful and the 29 remaining planned patients will be accrued. DLT for this study is defined as the occurrence of a severe adverse event (AE) that is at least possibly related to pembrolizumab, and occurs from the initiation of treatment thru 30 days after the final administration of the study treatment
Time Frame: Up to 20 weeks post treatment
Population: Participants enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Post Operative Radiotherapy
Number analyzed (Participants) | 18
Participants | 0

2. Primary Outcome: Number of Participants With Progression Free Survival
Description: Progression-free survival (PFS) will be calculated from treatment initiation to disease progression or death from any cause or last follow up
Time Frame: Up to 1 year after beginning treatment
Population: Participants enrolled in the study, excluding one participant who had disease progression prior to completing treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Post Operative Radiotherapy
Number analyzed (Participants) | 18
Participants | 17

ADVERSE EVENTS:
Time Frame: Up to 4 weeks after the last dose of trial treatment
Arm/Group | Pembrolizumab + Post Operative Radiotherapy
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Post Operative Radiotherapy (N=18)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Post Operative Radiotherapy (N=18)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Palpitations (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 5 (5)
Dry eye (Eye disorders) | 1 (2)
Subjunctival hemorrhage (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 10 (15)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Esophageal pain (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 6 (10)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Edema face (General disorders) | 1 (1)
Fatigue (General disorders) | 13 (24)
Fever (General disorders) | 1 (2)
Neck edema (General disorders) | 2 (2)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (2)
Otitis externa (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 15 (35)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (6)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 14 (30)
Platelet count decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 7 (14)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (16)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 14 (24)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
verrucas lesion ~1cm behind left ear (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT03057613/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT03057613/ICF_001.pdf